CLINICAL TRIAL: NCT02665598
Title: Prognostic Observation of Posterior Reversible Encephalopathy Syndrome
Acronym: POPRES
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yantai Yuhuangding Hospital (Other)
Collaborators: University of Southern California (Other)
Responsible Party: Sponsor
Other Study IDs: BoGao
Record Dates: First submitted 2016-01-03; First posted 2016-01-28 (Estimated); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Posterior Reversible Encephalopathy Syndrome
Keywords: Posterior Reversible Encephalopathy Syndrome,Prognosis
MeSH Terms: conditions — Posterior Leukoencephalopathy Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Posterior Reversible Encephalopathy Syndrome (PRES) is a clinical-radiological entity, which is associated with a variety of clinical conditions. The imaging and clinical findings are typically reversible, but many patients still have permanent neurological sequelae with a fatal outcome. Up to now there are no consistent conclusions about the factors that affecting its prognosis. The objective of our study is to discuss the effects of different causes, different imaging findings and laboratory parameters on the prognosis of PRES and deepen the understanding of the nature of PRES. This will contribute to predict the prognosis of patients with PRES and to further investigate the pathogenesis of PRES so as to guide the clinical treatment and follow-up evaluation. A multi-center retrospective case study will be performed from January 2016 to July 2017 and a total of 400 patients who meet the criteria for PRES diagnosis from 10 sub-centers are anticipated included in this research. Patients will be divided into several subgroups according to the etiology. Date will be collected from the clinical records，imaging and laboratory data of the patients, including demographic data, clinical data, imaging findings, laboratory parameters and follow-up data. During the follow-up, MRI and blood biochemical examination will be performed once more. The imaging findings of the patients will be assessed by two neuroimaging physicians, any difference between them will be agreed upon by consensus. Prognosis of the patients will be assessed by using the modified Rankin scale (mRS) scores. All of the above data is saved into the database. In this study we will review etiologies and imaging findings, laboratory and follow-up data of the patients we selected. Univariate and multivariate analysis will be performed within the group and between groups according to the subgroups. Then we will discuss the connection between different causes, different imaging findings and laboratory parameters and the prognosis of posterior reversible encephalopathy syndrome.

DETAILED DESCRIPTION:
Background and Significance

Posterior Reversible Encephalopathy Syndrome (PRES) is a clinical-radiological syndrome. It was first described by Hinchey et al. in 1996. It is characterized by a variable combination of headaches, seizures, altered mental status, visual impairment, nausea, vomiting and focal neurological signs and accompanied with symmetric vasogenic edema of bilateral posterior cerebral circulation territory. PRES is associated with multiple risk factors, such as renal dysfunction, hypertension, cytotoxic drugs, autoimmune disease and pre-eclampsia or eclampsia, which can occur in a wide range of diseases and predisposing factors. Lesions are usually located in the parietal occipital region. However, lesions may also involve unilateral cerebral hemisphere, anterior circulation area or deep brain structure. According to the location of the lesions, five distribution patterns were described: mainly parietal-occipital pattern, superior frontal sulcus pattern, holo-hemispheric watershed pattern, partial or asymmetric expression of the primary patterns and central pattern. In addition, cytotoxic edema with associated diffusion restriction, abnormal enhancement due to blood brain barrier disruption, hemorrhages, infarction are atypical findings which may be occasionally detected.

PRES is associated with a variety of clinical conditions. The occurrence of PRES is not affected by age and gender, it may present in all age groups. The occurrence of PRES may be a result of either breakdown of cerebral autoregulation and disruption of blood brain barrier, causing vasogenic edema or endothelial dysfunction resulting from circulating toxic mediators, sepsis, autoimmune conditions, or eclampsia. Up to now, the pathophysiological mechanism of PRES is still not clear, but cerebral autoregulation impairment and endothelial dysfunction are considered to be the most important potential mechanisms.

PRES usually has a favourable prognosis. The clinical and imaging findings are often reversible when the underlying causes are eliminated and the blood pressure is controlled. Even so, many patients still have permanent neurological sequelae and have a mortality of 5%-15%. Known risk factors for PRES include hypertension, renal disease and immunosuppressive therapy, and researchers have also found that lymphopenia and dyslipidemia are the potential risk factors for PRES. The prognostic factors of PRES include the presence of PRES risk factors, duration of symptoms, the presence of cytotoxic edema and hemorrhage. Alhilali et al. through the retrospective analysis of the etiologies, imaging findings and cerebrospinal fluid examination of the 47 PRES patients with lumbar puncture showed that clinical factors, imaging findings, cerebrospinal fluid laboratory results all affect the prognosis of PRES, with low CSF glucose, hypertensive encephalopathy, and imaging findings of hemorrhage increasing the risk of fatal outcome, while toxemia of pregnancy was found to have a relatively protective effect. Recent research had shown correlation of MRI findings and LDH and albumin levels, suggesting that these biochemical indices may be used as a prognostic factor. Although the various risk factors of PRES and its related imaging findings are well described, and in previous studies, the relationship between clinical factors, imaging findings, laboratory examination results and prognosis of PRES were analyzed respectively by different investigators, their relative effects on the prognosis are remain unclear and there are no consistent conclusions about it.

Here we use a multi-center approach to conduct this study to ensure a larger patients sample. This proposed multi-center retrospective study will analyze the factors that influence the prognosis of the patients with PRES. The aim of our research is to study the connection between different causes, different imaging findings, laboratory findings and clinical outcome in patients with PRES and deepen the understanding of the nature of PRES. The pathogenesis of PRES will be further discussed based on the results obtained. This will contribute to predict the prognosis of patients with PRES and to further investigate the pathogenesis of PRES so as to guide the clinical treatment and follow-up evaluation.

Research Design and Methods

1. Overall Design of The Research

   A multi-center retrospective case study, after securing required Institutional Review Board approval, will be performed from January 2016 to July 2015 and the patients with complete inpatient clinical records who meet the criteria from 10 sub-centers will be included. Patients' demographic data, clinical data, auxiliary examination, imaging findings and follow-up data will be collected and summarized. The imaging findings of the patients will be assessed by two neuroimaging physicians, any difference between them will be agreed upon by consensus. Following this, the connection between the different causes, different imaging findings, laboratory findings and clinical outcome of posterior reversible encephalopathy syndrome will be analyzed.
2. Patients and Grouping

   A total of 400 patients with complete inpatient clinical records who meet the criteria from 10 sub-centers will be included in this research. The patients above will be divided into several subgroups according to the causes of the disease, including hypertensive encephalopathy, cytotoxic drugs, toxemia of pregnancy (pre-eclampsia or eclampsia), autoimmune diseases and other diseases (anemia, hypomagnesemia, infection, sepsis, etc.).
3. Data Acquisition

   The following information will be collected by reviewing the medical records and follow-up of the patients who met the inclusion criteria:

   Basic information: demographic and sociological characteristics of patients, such as name, gender, age and so on; Clinical date: including the history of past illness, etiology, symptoms (headache, seizures, visual disturbances, nausea and vomiting, altered mental status, focal neurological signs, etc.), blood pressure/MAP at the time of attack, therapeutic measure, time from symptom onset to control of the causative factor, hospitalization, etc.

   Examination to identify cause of PRES: including blood biochemical examination (enzymes, metabolites, minerals, blood protein, etc.), lumbar puncture cerebrospinal fluid examination, EEG, blood gas analysis, etc.

   Imaging examination: including the time from PRES onset to MRI examination, location of lesion , the distribution pattern of edema, degree of edema, cytotoxic edema appears or not, abnormal enhanced appears or not, hemorrhage appears or not, MRA or DSA examination, perfusion weighted imaging, etc.

   Follow-up:

   Time interval from PRES onset to MRI follow-up; Follow up imaging findings; Prognosis observation: discharge status, including the partial or complete recovery of abnormal imaging, hemorrhagic and ischemic complications appear or not ,continue medication treatment or not (antihypertensive drugs, anticonvulsant drugs, etc.), death; time from symptoms onset to recovery of image abnormalities; recurrence and interval time; increased patient's current MRI and blood biochemical examination; the patients' mRS score at the time of onset, discharge and follow-up were achieved by review cases and follow-up.
4. Data Analysis

   All of the above data is saved into the database. In this study we will review etiologies and imaging findings, laboratory and follow-up data of the patients we selected. Univariate and multivariate analysis will be performed within the group and between groups according to the subgroups. In this research prognosis of the patients will be assessed by using the modified Rankin scale (mRS) scores. Single PRES related factors will be tested with Chi-square test. Intergroup comparison will be performed by using student t-test for normally distributed variables and Mann-Whitney U test for variables not normally distributed. In binary variable analysis, logistic regression analysis will be used to analysis factors related PRES. In polytomous variable analysis, multivariate logistic regression analysis will be performed to analyze factors related to PRES.
5. Quality Control

The patients will be identified strictly in accordance with the established inclusion and exclusion criteria. The imaging findings of the patients will be assessed by 2 neuroimaging physicians and the consensus will be reached through consultation when there were differences. The members of the group who assess the prognosis of PRES should be unified training.

Timeline of Events

Patients screening and data acquisition phase. The project is scheduled to initiate in April 2016 and complete all data collection in July 2016.

Data analysis phase. We plan to complete the data analysis in about 4 months after the data acquisition is completed.

Paper publishing stage. We plan to complete the paper publishing in about 6 months after the data analysis is finished.

Data opening phase. We plan to open the data to the society in stages after paper publishing is completed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who meet the criteria for PRES diagnosis:(1)typical symptoms and signs consistent with PRES, such as headache, seizures, mental status changes, visual disturbances or focal neurological deficits;(2)patients with typical or atypical imaging manifestations of PRES;(3)patients who have known risk factors of PRES.
2. Patients with definite prognosis will be included.
3. Patients with complete inpatient medical records will be included.

Exclusion Criteria:

1. Patients with edema secondary to ischemia, hemorrhage, infection, inflammation, or space occupying lesions will be excluded.
2. Patients with absent or non-diagnostic MRI will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients with complete inpatient clinical records who meet the inclusion criteria from January 2016 to July 2015 will be included in this research.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2016-04; Primary Completion 2023-07 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Quantitative assessment of short term and long term prognosis of PRES patients by mRS score | within six months

CONTACTS AND LOCATIONS:
Overall Officials: Bo Gao, MD, Study Chair
Locations (1):
- Weihai Municipal Hospital, Weihai, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Alhilali LM, Reynolds AR, Fakhran S. A multi-disciplinary model of risk factors for fatal outcome in posterior reversible encephalopathy syndrome. J Neurol Sci. 2014 Dec 15;347(1-2):59-65. doi: 10.1016/j.jns.2014.09.019. Epub 2014 Sep 22. PMID 25271189
- [Result] Merayo-Chalico J, Apodaca E, Barrera-Vargas A, Alcocer-Varela J, Colunga-Pedraza I, Gonzalez-Patino A, Arauz A, Abud-Mendoza C, Martinez-Martinez M, Gomez-Martin D. Clinical outcomes and risk factors for posterior reversible encephalopathy syndrome in systemic lupus erythematosus: a multicentric case-control study. J Neurol Neurosurg Psychiatry. 2016 Mar;87(3):287-94. doi: 10.1136/jnnp-2014-310145. Epub 2015 Mar 24. PMID 25804426
- [Result] Legriel S, Schraub O, Azoulay E, Hantson P, Magalhaes E, Coquet I, Bretonniere C, Gilhodes O, Anguel N, Megarbane B, Benayoun L, Schnell D, Plantefeve G, Charpentier J, Argaud L, Mourvillier B, Galbois A, Chalumeau-Lemoine L, Rivoal M, Durand F, Geffroy A, Simon M, Stoclin A, Pallot JL, Arbelot C, Nyunga M, Lesieur O, Troche G, Bruneel F, Cordoliani YS, Bedos JP, Pico F; Critically III Posterior Reversible Encephalopathy Syndrome Study Group (CYPRESS). Determinants of recovery from severe posterior reversible encephalopathy syndrome. PLoS One. 2012;7(9):e44534. doi: 10.1371/journal.pone.0044534. Epub 2012 Sep 14. PMID 23024751
- [Result] Liman TG, Bohner G, Endres M, Siebert E. Discharge status and in-hospital mortality in posterior reversible encephalopathy syndrome. Acta Neurol Scand. 2014 Jul;130(1):34-9. doi: 10.1111/ane.12213. Epub 2013 Dec 13. PMID 24329761
- [Result] Moon SN, Jeon SJ, Choi SS, Song CJ, Chung GH, Yu IK, Kim DH. Can clinical and MRI findings predict the prognosis of variant and classical type of posterior reversible encephalopathy syndrome (PRES)? Acta Radiol. 2013 Dec;54(10):1182-90. doi: 10.1177/0284185113491252. Epub 2013 Jul 15. PMID 23858507
- [Result] Pande AR, Ando K, Ishikura R, Nagami Y, Takada Y, Wada A, Watanabe Y, Miki Y, Uchino A, Nakao N. Clinicoradiological factors influencing the reversibility of posterior reversible encephalopathy syndrome: a multicenter study. Radiat Med. 2006 Dec;24(10):659-68. doi: 10.1007/s11604-006-0086-2. Epub 2006 Dec 25. PMID 17186320
- [Result] Pereira PR, Pinho J, Rodrigues M, Rocha J, Sousa F, Amorim J, Ribeiro M, Rocha J, Ferreira C. Clinical, imagiological and etiological spectrum of posterior reversible encephalopathy syndrome. Arq Neuropsiquiatr. 2015 Jan;73(1):36-40. doi: 10.1590/0004-282X20140176. Epub 2015 Jan 1. PMID 25608125
- [Result] Prasad N, Gulati S, Gupta RK, Kumar R, Sharma K, Sharma RK. Is reversible posterior leukoencephalopathy with severe hypertension completely reversible in all patients? Pediatr Nephrol. 2003 Nov;18(11):1161-6. doi: 10.1007/s00467-003-1243-9. Epub 2003 Sep 19. PMID 14505162
- [Result] Singh RR, Ozyilmaz N, Waller S, U-King-Im JM, Lim M, Siddiqui A, Sinha MD. A study on clinical and radiological features and outcome in patients with posterior reversible encephalopathy syndrome (PRES). Eur J Pediatr. 2014 Sep;173(9):1225-31. doi: 10.1007/s00431-014-2301-y. Epub 2014 Apr 16. PMID 24737291
- [Result] Postma IR, Slager S, Kremer HP, de Groot JC, Zeeman GG. Long-term consequences of the posterior reversible encephalopathy syndrome in eclampsia and preeclampsia: a review of the obstetric and nonobstetric literature. Obstet Gynecol Surv. 2014 May;69(5):287-300. doi: 10.1097/OGX.0000000000000069. PMID 25101694
- [Result] Liman TG, Bohner G, Heuschmann PU, Endres M, Siebert E. The clinical and radiological spectrum of posterior reversible encephalopathy syndrome: the retrospective Berlin PRES study. J Neurol. 2012 Jan;259(1):155-64. doi: 10.1007/s00415-011-6152-4. Epub 2011 Jun 30. PMID 21717193
- [Result] Fugate JE, Rabinstein AA. Posterior reversible encephalopathy syndrome: clinical and radiological manifestations, pathophysiology, and outstanding questions. Lancet Neurol. 2015 Sep;14(9):914-925. doi: 10.1016/S1474-4422(15)00111-8. Epub 2015 Jul 13. PMID 26184985
- [Result] Gao B, Liu FL, Zhao B. Association of degree and type of edema in posterior reversible encephalopathy syndrome with serum lactate dehydrogenase level: initial experience. Eur J Radiol. 2012 Oct;81(10):2844-7. doi: 10.1016/j.ejrad.2011.12.010. Epub 2011 Dec 29. PMID 22209526
- [Result] Gao B, Yu BX, Li RS, Zhang G, Xie HZ, Liu FL, Lv C. Cytotoxic Edema in Posterior Reversible Encephalopathy Syndrome: Correlation of MRI Features with Serum Albumin Levels. AJNR Am J Neuroradiol. 2015 Oct;36(10):1884-9. doi: 10.3174/ajnr.A4379. Epub 2015 Jul 2. PMID 26138140
- [Result] Bo G, Hui L, Feng-Li L, Cui L. Relationships between edema degree and clinical and biochemical parameters in posterior reversible encephalopathy syndrome: a preliminary study. Acta Neurol Belg. 2012 Sep;112(3):281-5. doi: 10.1007/s13760-012-0060-y. Epub 2012 Mar 24. PMID 22450710